CLINICAL TRIAL: NCT03647059
Title: Real-time Noninvasive Assessment of Donor Liver Quality
Brief Title: Rapid Assessment of Donor Liver Quality
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Lin Zhong, Director of hepatobiliary surgery, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Other Study IDs: SHLTQC-2
Record Dates: First submitted 2018-08-09; First posted 2018-08-27 (Actual); Last update posted 2018-08-27 (Actual); Status verified 2018-08

CONDITIONS: Transplant; Failure, Liver

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Biospecimen Retention: Samples Without DNA — we just need to cut a little piece of donor liver to conduct a examination of Laser scanning Confocal Microscopy(LSCM)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- LSCM examination
  Interventions: Diagnostic Test: LSCM examination

INTERVENTIONS:
Diagnostic Test: LSCM examination — Cut a piece of donor liver and conduct the LSCM examination after staining fluorescein

SUMMARY:
Aims：

1. Conduct multi-center, prospective and open research on liver quality assessment and establish LSCM liver quality assessment system
2. Classification of liver quality grades by LSCM for different pathological conditions (steatosis, fibrosis, hepatocyte necrosis, etc.)
3. Compare the specificity and sensitivity of LSCM evaluation results with the results of liver donor quality evaluation and intraoperative pathological biopsy results.
4. LSCM classifies the quality of donor liver and compares the recovery of liver function on the first day after liver transplantation.
5. LSCM grades the quality of donor liver and compares the long-term prognosis

ELIGIBILITY:
Inclusion Criteria:

* All donor livers to be used for liver transplantations

Exclusion Criteria:

* Exclusion of multiple organ transplantation
* Exclusion of detached transplantation and partial liver transplantation, etc.
* Removal of blood type incompatible patients for transplantation
* Exclusion of poor donor liver quality due to surgical technique (such as hepatic artery embolization) , portal vein thrombosis, etc.)
* Any form of substance abuse, mental illness or any disease that the investigator believes may interfere with the patient's understanding of the research requirements.
* Can not complete routine research follow-up, and other circumstances that the investigator believes are not suitable for the experiment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All donor livers to be used for liver transplantations. Before transplant, the donor liver will be stored in the cold-UW solution in ice water. We just cut a piece of liver simple in the any place of donor liver, usually, we always cut a piece of liver simple from the edge of the donor liver.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2018-08-15 (Estimated); Primary Completion 2020-08-15 (Estimated); Study Completion 2022-08-15 (Estimated)

PRIMARY OUTCOMES:
LSCM examination results | 1 day
  LSCM examination is focus on the detections of the hepatocyte nucleus and the micro structures(such as the micro-circulation、central vein and so on).

SECONDARY OUTCOMES:
HE section staining pathological examination | 1 week
  All of donor livers must be detected by HE section staining pathological examination and it is mainly focused on the detection of hepatocyte nucleus and the micro structures(such as the micro-circulation、central vein and so on).

OTHER OUTCOMES:
Clinical examinations | 1 week
  Mainly focus on the examinations such as ALT、AST、LDH and so on.

CONTACTS AND LOCATIONS:
Overall Officials: Zhong Lin, doctor, Principal Investigator — Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, China
Locations (1):
- Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
positive IPD is available to other researchers
Supporting Information: Study Protocol